CLINICAL TRIAL: NCT00110084
Title: Phase II Trial of Weekly Nab (Nanoparticle Albumin Bound)-Paclitaxel (Nab-paclitaxel) (Abraxane®) in Combination With Gemcitabine in Patients With Metastatic Breast Cancer
Brief Title: ABI-007 (Nab-Paclitaxel) and Gemcitabine in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Vivek Roy, M.D., Mayo Clinic Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000423195; U10CA025224 (NIH); N0531 (Other: Mayo Clinic Cancer Cancer and NCCTG); 855-05 (Other: Mayo Clinic IRB); N0433 (Other: NCCTG Old Protocol)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Results first posted 2011-05-26 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nab-paclitaxel/Gemcitabine (Experimental)
  Interventions: Drug: Gemcitabine; Drug: Paclitaxel protein-bound particles for injectable suspension (albumin-bound)

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m2 (IV over 30 min) (days 1 and 8) on 21 day cycle
  Other Names: Gemzar
Drug: Paclitaxel protein-bound particles for injectable suspension (albumin-bound) — 125 mg/m2 (IV over 30 min) (days 1 and 8) on 21 day cycle
  Other Names: nab (nanoparticle albumin-bound)-Paclitaxel, Abraxane

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ABI-007(Nab-Paclitaxel((Nanoparticle Albumin Bound)-Paclitaxel)) and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving ABI-007 together with gemcitabine works in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of ABI-007 and gemcitabine, in terms of response rate in women with metastatic breast cancer.
* Determine the toxicity profile of this regimen, in terms of incidence and severity of observed toxic effects, in these patients.

Secondary

* Determine the time to disease progression and survival of patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive ABI-007 IV over 30 minutes and gemcitabine IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for up to 5 years.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed invasive breast cancer

  - Clinical evidence of metastatic disease

  + No bone metastases or other non-measurable disease as the only evidence of metastasis
* Measurable disease, defined as at least 1 measurable lesion

  - The following are considered non-measurable disease:
  * Small lesions (< 2 cm)
  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural or pericardial effusions
  * Inflammatory breast disease
  * Lymphangitis cutis or pulmonis
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions
* HER2(human epidermal growth factor receptor 2)-positive disease allowed provided patient has received prior treatment with trastuzumab
* No evidence of active brain metastasis, including leptomeningeal involvement
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over Sex
* Female Menopausal status
* Not specified Performance status
* ECOG 0-1 Life expectancy
* At least 12 weeks Hematopoietic
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL Hepatic
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN Renal
* Creatinine ≤ 1.5 mg/dL Other
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after completion of study treatment
* No pre-existing peripheral neuropathy > grade 1
* No other clinically significant illness or significant medical condition that would preclude study participation
* No history of allergy or hypersensitivity to paclitaxel protein-bound particles in an injectable suspension, paclitaxel, gemcitabine, albumin, drug product excipients, or agents that are chemically similar to study drugs
* No serious medical risk factors involving any of the major organ systems that would preclude study participation
* No active stage III or IV invasive non-breast malignancy within the past 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics Chemotherapy
* No more than 1 prior adjuvant chemotherapy regimen
* No prior chemotherapy for metastatic disease
* At least 6 months since prior adjuvant or neoadjuvant taxane
* More than 2 weeks since prior cytotoxic chemotherapy
* Prior neoadjuvant chemotherapy allowed
* No other concurrent chemotherapy Endocrine therapy
* Prior hormonal treatment as adjuvant therapy or for metastatic disease allowed Radiotherapy
* Prior radiotherapy to target lesion allowed provided there is evidence of disease progression after completion of treatment
* More than 2 weeks since prior radiotherapy, except radiotherapy to a non-target lesion only or single-dose palliative radiotherapy
* No concurrent radiotherapy Surgery
* Not specified Other
* More than 2 weeks since prior investigational drugs
* No concurrent participation in another clinical trial that is studying investigational procedures or therapies
* Concurrent bisphosphonates (e.g., pamidronate or zoledronate) allowed for palliation of pain or lytic lesions from breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-08; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Roy, MD, FACP, Study Chair — Mayo Clinic; Philip J. Stella, MD, Study Chair — CCOP - Michigan Cancer Research Consortium; Tom R. Fitch, M.D., Principal Investigator — Mayo Clinic; Timothy J. Hobday, M.D., Principal Investigator — Mayo Clinic
Locations (201):
- United States (201):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thorton, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Cancer Research Center of Hawaii, Honolula, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - St. Francis Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, P. C., Ames, Iowa
  - Bettendorf, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center Cancer Center, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, P.A. - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, P.A. - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, P.A. - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, P.A. - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, P.A. - Salina, Salina, Kansas
  - Cancer Center of Kansas, P.A. - Wellington, Wellington, Kansas
  - Associates in Womens Health, P.A. - North Review, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, P.C., Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - Immanuel St. Joseph's Clinic, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Toledo Surgical Specialists, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - United States Air Force Medical Center Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Result] Roy V, LaPlant BR, Gross GG, Bane CL, Palmieri FM; North Central Cancer Treatment Group. Phase II trial of weekly nab (nanoparticle albumin-bound)-paclitaxel (nab-paclitaxel) (Abraxane) in combination with gemcitabine in patients with metastatic breast cancer (N0531). Ann Oncol. 2009 Mar;20(3):449-53. doi: 10.1093/annonc/mdn661. Epub 2008 Dec 15. PMID 19087987
- [Result] Roy V, LaPlant BR, Gross GG, et al.: NCCTG phase II trial N0531of weekly nab-paclitaxel (nab-p) in combination with gemcitabine (gem) in patients with metastatic breast cancer (MBC). [Abstract] J Clin Oncol 25 (Suppl 18): A-1048, 2007.
- [Result] Moreno-Aspitia A, Perez EA. North Central Cancer Treatment Group N0531: Phase II Trial of weekly albumin-bound paclitaxel (ABI-007; Abraxane) in combination with gemcitabine in patients with metastatic breast cancer. Clin Breast Cancer. 2005 Oct;6(4):361-4. doi: 10.3816/CBC.2005.n.042. No abstract available. PMID 16277889

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 22 medical clinics in the United States between November 2005 to May 2006
Groups:
- Nab-paclitaxel/Gemcitabine: Nab (nanoparticle albumin-bound)-Paclitaxel (125mg/m^2)(IV over 30 min) (days 1 and 8) on 21 day cycle and gemcitabine (1000 mg/m^2)(IV over 30 min) (days 1 and 8) on 21 day cycle
Period: Overall Study
Arm/Group | Nab-paclitaxel/Gemcitabine
Started | 50
Completed | 22
Not Completed | 28
Not completed — Adverse Event | 9
Not completed — Death | 1
Not completed — Patient Refusal | 10
Not completed — Alternate Therapy | 5
Not completed — Intercurrent Illness | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nab-paclitaxel/Gemcitabine
Number analyzed (Participants) | 50
Age Continuous [Median (Full Range); unit: years] | 56 [29 to 86]
Sex/Gender, Customized [Number; unit: participants]
  Female | 50
Region of Enrollment [Number; unit: participants]
  United States | 50
Dominant disease site [Number; unit: participants]
  Soft tissue | 5
  Osseous | 4
  Visceral | 41
Estrogen receptor status [Number; unit: participants] — Using IHC (Immunohistochemistry): categorization is determined by individual institution standards.
  participants
    Positive | 34
    Negative | 14
    Unknown | 2
HER2 (human epidermal growth factor receptor 2) status [Number; unit: participants]
  Positive | 1
  Negative | 49
Number of metastatic sites [Number; unit: participants]
  1 | 5
  2 | 15
  3+ | 30
Performance Score [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  participants
    0 - Fully Active | 23
    1 - Ambulatory, restricted strenuous activity | 27
Progesterone receptor status [Number; unit: participants] — Using IHC (Immunohistochemistry): categorization is determined by individual institution standards.
  participants
    Positive | 28
    Negative | 20
    Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Confirmed Responses
Description: Confirmed tumor response (complete and partial) as measured by RECIST(Response Evaluation Criteria In Solid Tumors) criteria on 2 consecutive evaluations at least 6 weeks apart.
  Confirmed tumor response is at least a 30% decrease in the sum of the longest diameter of target lesions and no new lesions.
Time Frame: Two consecutive evaluations at least 6 weeks apart
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Nab-paclitaxel/Gemcitabine
Number analyzed (Participants) | 50
participants
  Confirmed response | 25
  Assessable | 50
Statistical Analysis 1: Comparison: Nab-paclitaxel/Gemcitabine; Proportion of confirmed responses was estimated by the number of patients who achieved a confirmed response divided by the total number of assessable patients; Test type: Superiority or Other; Proportion of confirmed responses (%) = 50, 95% CI 2-sided [36 to 64] — 95% Confidence intervals were calculated for the true confirmed response rate using properties of the binomial distribution

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the number of months from registration to the date of disease progression or death, with patients who are alive and progression free being censored on the date of their last evaluation.
Time Frame: Time from registration to progression or death (up to 5 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel/Gemcitabine
Number analyzed (Participants) | 50
months | 7.9 [5.4 to 10]

3. Secondary Outcome: Overall Survival
Description: Overall survival time was defined as the number of days from registration to the date of death or last follow-up
Time Frame: Death or last follow-up (up to 5 years)
Population: Median survival time from Kaplan-meir estimate has not been attained.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel/Gemcitabine
Number analyzed (Participants) | 0

4. Secondary Outcome: Adverse Event
Description: Number of patients that experienced adverse events (grade 3 or more occurring in >5% of patients) as measured by NCI CTCAE (Common Terminology Criteria for Adverse Events) v3.0
Time Frame: Every 6 weeks
Measure: Number; unit: participants
Arm/Group | Nab-paclitaxel/Gemcitabine
Number analyzed (Participants) | 50
participants
  Neutropenia | 27
  Fatigue | 14
  Anemia | 7
  Dyspnea | 7
  Thrombocytopenia | 6
  Arthralgia | 4
  Vomiting | 4
  Neuropathy | 3
  Myalgia | 3
  Nausea | 3
  Pain-abdominal | 3
  Aspartate aminotransferase (AST) | 3

ADVERSE EVENTS:
Arm/Group | Nab-paclitaxel/Gemcitabine
Serious Adverse Events (participants affected / at risk) | 11/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-paclitaxel/Gemcitabine (N=50)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Arrythmia (Cardiac disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain-Abdominal (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Neutropenia (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-paclitaxel/Gemcitabine (N=50)
Anemia (Blood and lymphatic system disorders) | 47 (302)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Vision-Blurred (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea-No Colostom (Gastrointestinal disorders) | 18 (33)
Nausea (Gastrointestinal disorders) | 30 (101)
Oral cavity Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 1 (1)
Oral cavity Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 18 (35)
Pain-Abdominal (Gastrointestinal disorders) | 4 (7)
Pain-Stomach (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 18 (34)
Edema: Head/Neck (General disorders) | 1 (1)
Edema: Limb (General disorders) | 8 (14)
Edema: trunk/genital (General disorders) | 1 (1)
Fatigue (General disorders) | 48 (269)
Fever-No ANC (General disorders) | 16 (26)
Pain (General disorders) | 3 (3)
Hypersensitivity (Immune system disorders) | 1 (1)
Bladder infection (Infections and infestations) | 3 (3)
Bronchial infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 3 (5)
Lung (pneumonia) infection (Infections and infestations) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus infection (Infections and infestations) | 1 (2)
Skin (cellulites) infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 7 (14)
Alkaline phosphatase (Investigations) | 2 (5)
Amylase (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (12)
Blood bilirubin increased (Investigations) | 1 (1)
Leukopenia (Investigations) | 10 (16)
Lipase increased (Investigations) | 1 (5)
Lymphopenia (Investigations) | 1 (1)
Metabolic/Lab (Investigations) | 1 (2)
Neutropenia (Investigations) | 44 (194)
Platelet count decreased (Investigations) | 40 (121)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (6)
Anorexia (Metabolism and nutrition disorders) | 5 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (21)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (5)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (117)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Extremity-lower weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 29 (94)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (3)
Headache (Nervous system disorders) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 26 (145)
Syncope (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 30 (115)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharynx Mucositis/stomatitis (functional/symptomatic) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 45 (304)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 5 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 4 (7)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (3)
Phlebitis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes